CLINICAL TRIAL: NCT05447000
Title: The Effect of Mindfulness-Based Practices and Deep Relaxation Exercises on Pregnancy-Related Anxiety Level
Brief Title: The Effect of Mindfulness-Based Practices and Deep Relaxation Exercises in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Assist. Prof. Dr. in the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya University
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Pregnancy Related
MeSH Terms: conditions — Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfullness Based Stress Reduction (Experimental): Mindfullness Based Stress Reduction (MBSR) therapy
  Interventions: Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention
- Deep Relaxation Exercises (Experimental): Deep Relaxation Exercises therapy
  Interventions: Behavioral: Deep Relaxation Exercises intervention
- Control (Other): Control
  Interventions: Other: No Intervention

INTERVENTIONS:
Behavioral: Mindfullness Based Stress Reduction (MBSR) intervention — Mindfullness Based Stress Reduction (MBSR) intervention: Monitoring anxiety levels with mindfulness program
  Arms: Mindfullness Based Stress Reduction
Behavioral: Deep Relaxation Exercises intervention — Deep Relaxation Exercises intervention: Monitoring anxiety levels with deep Relaxation Exercises intervention
  Arms: Deep Relaxation Exercises
Other: No Intervention — No Intervention
  Arms: Control

SUMMARY:
Pregnancy is a transitional period during which important physical, biological and psychological changes are experienced for women, and the probability of encountering factors that may cause stress, anxiety and low quality of life is high. Maternal stress in pregnancy is associated with negative birth outcomes and can be reduced with relaxation exercises. However, mindfulness-based approaches affect pregnancy outcomes positively. Data collected with the "Personal Description Form", and "The Pregnancy-related Anxiety Questionnaire-Revised 2".

DETAILED DESCRIPTION:
Pregnancy is a transitional period during which important physical, biological and psychological changes are experienced for women, and the probability of encountering factors that may cause stress, anxiety and low quality of life is high. Maternal stress in pregnancy is associated with negative birth outcomes and can be reduced with relaxation exercises. However, mindfulness-based approaches affect pregnancy outcomes positively. The aim of this study, which was conducted to determine the effects of mindfulness practices and deep relaxation exercises on the level of pregnancy-related anxiety, is to create intervention programs compatible with the prenatal period and to contribute to the improvement of pregnancy outcomes. First of all, a total of 111 pregnant women (37 mindfulness based stress reduction program, 37 deep relaxation exercises and 37 control) are planned to be included in the study. However, we recalculated the power analysis with a reference study after obtaining approval and before starting the study. With the calculation we made with the reference study, we determined our final sample number as 102 pregnant women (34 individuals for the mindfulness meditation group, 34 individuals for the deep relaxation exercises group, and 34 individuals for the control group). Data collected with the "Personal Description Form", and "The Pregnancy-related Anxiety Questionnaire-Revised 2". Mindfulness and deep relaxation practices was applied by midwives who are experts in their fields who are certified in these fields.

ELIGIBILITY:
Inclusion Criteria:

* Having internet access,
* Without any diagnosed psychiatric health problem,
* At 12-24 weeks of gestation,
* There is no risk factor in pregnancy,
* Literate,
* Using smart phone,
* Having a headset accessory for phone calls,
* Pregnant women who voluntarily agreed to participate in the study

Exclusion Criteria:

-Mental disabilities

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant
Enrollment: 95 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Scale | At the end of the 1 months
  For primiparas, a minimum of 11 points and a maximum of 55 points is obtained, and for multipars, a minimum of 10 and a maximum of 50 points are obtained. As the score obtained from the scale increases, it is accepted that the level of anxiety in pregnancy is higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gokbulut N, Cengizhan SO, Akca EI, Ceran E. The effects of a mindfulness-based stress reduction program and deep relaxation exercises on pregnancy-related anxiety levels: A randomized controlled trial. Int J Nurs Pract. 2024 Oct;30(5):e13238. doi: 10.1111/ijn.13238. Epub 2024 Jan 26. PMID 38279199